CLINICAL TRIAL: NCT03986996
Title: Antimicrobial Therapy for Ulcerative Colitis : Evaluation of Two Antibiotic Combinations for Refractory Ulcerative Colitis
Brief Title: Antimicrobial Therapy for Ulcerative Colitis (UC)
Acronym: UC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: There is no feasibility to conduct the study
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Arie Levine, Director, Pediatric Gastroenterology and Nutrition Unit, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AntimicrobialUC
Record Dates: First submitted 2019-06-04; First posted 2019-06-14 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Amoxicillin; Metronidazole; Doxycycline

STUDY DESIGN:
Intervention Model Description: 2 groups with 1:1 randomization
Who Masked: Investigator
Masking Description: The investigator will be blinded to the study group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 -Amoxycillin Doxycyclin and metronidazole (Active Comparator): triple therapy with amoxicillin, metronidazole and tetracycline twice daily, for 2 weeks.
  Interventions: Drug: amoxicillin, metronidazole and doxycycline
- Group 2 -Amoxycillin and Doxycyclin (Experimental): double therapy with Amoxycillin and Doxycyclin twice daily, for 2 weeks.
  Interventions: Drug: amoxicillin and doxycyclin

INTERVENTIONS:
Drug: amoxicillin, metronidazole and doxycycline — antibiotics: Patient weight 30-50 kg Patient weight > 50 kg Tetracycline 50 mg X 2 Day X 2 weeks 100 mg X 2 Day X 2 weeks Amoxicillin 750 mg X 2 Day X 2 weeks 750 mg X 2 Day X 2 weeks Metronidazole 250 mg X 2 Day X 2 weeks 375 mg X 2 Day X 2 weeks
  Other Names: Amoxy, Flagyl, Doxylin
  Arms: Group 1 -Amoxycillin Doxycyclin and metronidazole
Drug: amoxicillin and doxycyclin — antibiotics: Patient weight 30-50 kg Patient weight > 50 kg Tetracycline 50 mg X 2 Day X 2 weeks 100 mg X 2 Day X 2 weeks Amoxicillin 750 mg X 2 Day X 2 weeks 750 mg X 2 Day X 2 weeks
  Other Names: Amoxy, Doxylin
  Arms: Group 2 -Amoxycillin and Doxycyclin

SUMMARY:
The Aim of this randoized controlled pilot study is to find a better treatment strategy for active UC based on the recent knowledge regarding the microbiota in UC and the beneficial or detrimental effects of antibiotics in restoring gut health and reducing inflammation. This study is designed to determine whether therapy with two antibiotics during a flare - amoxicillin and doxycillin, will be better than the current published antibiotic treatment combination using these antibiotics with metronidazole ( as the latter which may degrade beneficial species without adding benefit towards reducing pathobionts)

DETAILED DESCRIPTION:
Recent studies suggest that UC is associated with alterations of the microbiota. Further support for targeting the microbiota includes several studies demonstrating that antibiotics might be helpful for severe refractory colitis. Antibiotics may work by reducing pathobionts, by causing niche expansion of beneficial bacteria , and may harm if they do not reduce pathobionts or reduce beneficial commensals Recently, a triple antibiotic therapy with amoxicillin, metronidazole and tetracycline was developed for UC. However, a recent study on the effect of 11 different oral antibiotics on gut bacteria found that seven of them including metronidazole might cause lbacterial translocation . Anaerobes are critical for butyrate production. .

Based on these recent studies, it would appear that tetracycline and amoxicillin are more likely to cause the beneficial effect, while metronidazole might actually be detrimental. Thus by removing metronidazole the investigators might actually have a better effect both for efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of UC, disease confined to the large intestine, involving the rectosigmoid for at least 3 months.
2. Weight >30 kg
3. Mild to Moderate active disease, SCCAI of ≥5 and ≤ 10, 10 ≤ PUCAI ≤4.
4. Refractory to mesalamine 6 weeks, or steroids > 14 days, or immunomodulator 12 weeks or biologics at least 12 weeks therapy.

Exclusion Criteria:

1. Start of a new biologic in the previous 12 weeks.
2. Proctitis
3. Evidence for Clostridium difficile infection.
4. Any proven current infection such as CMV, positive stool culture or parasite.
5. Current Extra intestinal manifestation of UC such as active arthritis or PSC.
6. Immune deficiency (other than drug induced).
7. Current use of a calcineurin inhibitor
8. Pregnancy.
9. Suspected toxic megacolon, guarding on palpation, or signs of peritoneal inflammation
10. Patients with other IBD unrelated disease such as autoimmune disorders, renal failure, fever or current infection (UTI, strep throat, pneumonia, etc), prior or current neoplasia
11. Fever >38
12. Participation in another clinical interventional trial
13. An active malignant disease or a prior malignancy during the previous 5 years (excluding skin BCC).
14. Anticipation for antibiotic use within the study period (such as for elective surgery or dental treatment).
15. Acute severe UC in the past 3 months.
16. Presence of a pouch or pouchitis.

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Efficacy - Clinical Response in group 1 and 2 or Clinical Remission | Week 3
  Response defined as a 3 point drop in SCCAI / 20 point drop in PUCAI or drop in less than 3/20 point but entering clinical remission, defined as a SCCAI score<5 / PUCAI score<10.
  Remission defined as SCCAI score<5 / PUCAI score<10.
  SCCAI - simple clinical colitis activity index. The calculated score ranges from 0 to 19, where active disease is a score of 5 or higher.
  PUCAI - pediatric Ulcerative colitis activity index. The calculated score ranges from 0 to 85, where active disease is a score of 10 or higher.

SECONDARY OUTCOMES:
Efficacy - Clinical Response in group 1 and 2 | Week 6
  Mean/median SCCAI / PUCAI
  SCCAI - simple clinical colitis activity index. The calculated score ranges from 0 to 19, where active disease is a score of 5 or higher.
  PUCAI - pediatric Ulcerative colitis activity index. The calculated score ranges from 0 to 85, where active disease is a score of 10 or higher.
EFFICACY - Remission | Week 6
  SCCAI score<5 / PUCAI score<10.
  SCCAI - simple clinical colitis activity index. The calculated score ranges from 0 to 19, where active disease is a score of 5 or higher.
  PUCAI - pediatric Ulcerative colitis activity index. The calculated score ranges from 0 to 85, where active disease is a score of 10 or higher.
EFFICACY - PGA | Week 6
  Physicians Global Assessment
  Values:
  1. Normal, not at all ill
  2. Borderline ill
  3. Mildly ill
  4. Moderately ill
  5. Markedly ill
  6. Severely ill
  7. Among the most extremely ill patients
EFFICACY - Corticosteroid free remission | Week 6
  Remission defined as SCCAI score<5 / PUCAI score<10.
  SCCAI - simple clinical colitis activity index. The calculated score ranges from 0 to 19, where active disease is a score of 5 or higher.
  PUCAI - pediatric Ulcerative colitis activity index. The calculated score ranges from 0 to 85, where active disease is a score of 10 or higher.
EFFICACY - Corticosteroid free remission | Week 12
  Remission defined as SCCAI score<5 / PUCAI score<10.
  SCCAI - simple clinical colitis activity index. The calculated score ranges from 0 to 19, where active disease is a score of 5 or higher.
  PUCAI - pediatric Ulcerative colitis activity index. The calculated score ranges from 0 to 85, where active disease is a score of 10 or higher.
EFFICACY - Decrease in endoscopic disease activity | Week 12
  Decrease in endoscopic disease activity mesured with the Simple Endoscopic Score for Crohn's Disease (SES-CD). The calculated score ranges from 0 to 60

CONTACTS AND LOCATIONS:
Overall Officials: Dror Weiner, MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- The E.Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jostins L, Ripke S, Weersma RK, Duerr RH, McGovern DP, Hui KY, Lee JC, Schumm LP, Sharma Y, Anderson CA, Essers J, Mitrovic M, Ning K, Cleynen I, Theatre E, Spain SL, Raychaudhuri S, Goyette P, Wei Z, Abraham C, Achkar JP, Ahmad T, Amininejad L, Ananthakrishnan AN, Andersen V, Andrews JM, Baidoo L, Balschun T, Bampton PA, Bitton A, Boucher G, Brand S, Buning C, Cohain A, Cichon S, D'Amato M, De Jong D, Devaney KL, Dubinsky M, Edwards C, Ellinghaus D, Ferguson LR, Franchimont D, Fransen K, Gearry R, Georges M, Gieger C, Glas J, Haritunians T, Hart A, Hawkey C, Hedl M, Hu X, Karlsen TH, Kupcinskas L, Kugathasan S, Latiano A, Laukens D, Lawrance IC, Lees CW, Louis E, Mahy G, Mansfield J, Morgan AR, Mowat C, Newman W, Palmieri O, Ponsioen CY, Potocnik U, Prescott NJ, Regueiro M, Rotter JI, Russell RK, Sanderson JD, Sans M, Satsangi J, Schreiber S, Simms LA, Sventoraityte J, Targan SR, Taylor KD, Tremelling M, Verspaget HW, De Vos M, Wijmenga C, Wilson DC, Winkelmann J, Xavier RJ, Zeissig S, Zhang B, Zhang CK, Zhao H; International IBD Genetics Consortium (IIBDGC); Silverberg MS, Annese V, Hakonarson H, Brant SR, Radford-Smith G, Mathew CG, Rioux JD, Schadt EE, Daly MJ, Franke A, Parkes M, Vermeire S, Barrett JC, Cho JH. Host-microbe interactions have shaped the genetic architecture of inflammatory bowel disease. Nature. 2012 Nov 1;491(7422):119-24. doi: 10.1038/nature11582. PMID 23128233
- [Background] Manichanh C, Borruel N, Casellas F, Guarner F. The gut microbiota in IBD. Nat Rev Gastroenterol Hepatol. 2012 Oct;9(10):599-608. doi: 10.1038/nrgastro.2012.152. Epub 2012 Aug 21. PMID 22907164
- [Background] Noor SO, Ridgway K, Scovell L, Kemsley EK, Lund EK, Jamieson C, Johnson IT, Narbad A. Ulcerative colitis and irritable bowel patients exhibit distinct abnormalities of the gut microbiota. BMC Gastroenterol. 2010 Nov 12;10:134. doi: 10.1186/1471-230X-10-134. PMID 21073731
- [Background] Davenport M, Poles J, Leung JM, Wolff MJ, Abidi WM, Ullman T, Mayer L, Cho I, Loke P. Metabolic alterations to the mucosal microbiota in inflammatory bowel disease. Inflamm Bowel Dis. 2014 Apr;20(4):723-31. doi: 10.1097/MIB.0000000000000011. PMID 24583479
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] James SL, Christophersen CT, Bird AR, Conlon MA, Rosella O, Gibson PR, Muir JG. Abnormal fibre usage in UC in remission. Gut. 2015 Apr;64(4):562-70. doi: 10.1136/gutjnl-2014-307198. Epub 2014 Jul 18. PMID 25037189
- [Background] Khalil NA, Walton GE, Gibson GR, Tuohy KM, Andrews SC. In vitro batch cultures of gut microbiota from healthy and ulcerative colitis (UC) subjects suggest that sulphate-reducing bacteria levels are raised in UC and by a protein-rich diet. Int J Food Sci Nutr. 2014 Feb;65(1):79-88. doi: 10.3109/09637486.2013.825700. Epub 2013 Aug 13. PMID 23941288
- [Background] De Preter V, Arijs I, Windey K, Vanhove W, Vermeire S, Schuit F, Rutgeerts P, Verbeke K. Decreased mucosal sulfide detoxification is related to an impaired butyrate oxidation in ulcerative colitis. Inflamm Bowel Dis. 2012 Dec;18(12):2371-80. doi: 10.1002/ibd.22949. Epub 2012 Mar 20. PMID 22434643
- [Background] Jowett SL, Seal CJ, Pearce MS, Phillips E, Gregory W, Barton JR, Welfare MR. Influence of dietary factors on the clinical course of ulcerative colitis: a prospective cohort study. Gut. 2004 Oct;53(10):1479-84. doi: 10.1136/gut.2003.024828. PMID 15361498
- [Background] Pitcher MC, Beatty ER, Cummings JH. The contribution of sulphate reducing bacteria and 5-aminosalicylic acid to faecal sulphide in patients with ulcerative colitis. Gut. 2000 Jan;46(1):64-72. doi: 10.1136/gut.46.1.64. PMID 10601057
- [Background] Ohkusa T, Nomura T, Terai T, Miwa H, Kobayashi O, Hojo M, Takei Y, Ogihara T, Hirai S, Okayasu I, Sato N. Effectiveness of antibiotic combination therapy in patients with active ulcerative colitis: a randomized, controlled pilot trial with long-term follow-up. Scand J Gastroenterol. 2005 Nov;40(11):1334-42. doi: 10.1080/00365520510023648. PMID 16334443
- [Background] Ohkusa T, Kato K, Terao S, Chiba T, Mabe K, Murakami K, Mizokami Y, Sugiyama T, Yanaka A, Takeuchi Y, Yamato S, Yokoyama T, Okayasu I, Watanabe S, Tajiri H, Sato N; Japan UC Antibiotic Therapy Study Group. Newly developed antibiotic combination therapy for ulcerative colitis: a double-blind placebo-controlled multicenter trial. Am J Gastroenterol. 2010 Aug;105(8):1820-9. doi: 10.1038/ajg.2010.84. Epub 2010 Mar 9. PMID 20216533
- [Background] Turner D, Levine A, Kolho KL, Shaoul R, Ledder O. Combination of oral antibiotics may be effective in severe pediatric ulcerative colitis: a preliminary report. J Crohns Colitis. 2014 Nov;8(11):1464-70. doi: 10.1016/j.crohns.2014.05.010. Epub 2014 Jun 20. PMID 24958064
- [Background] Terao S, Yamashiro K, Tamura I, Hirano T, Ohkusa T, Kato K. Antibiotic combination therapy for steroid withdrawal in steroid-dependent ulcerative colitis. Digestion. 2011;83(3):198-203. doi: 10.1159/000321811. Epub 2011 Jan 21. PMID 21266816
- [Background] Kato K, Ohkusa T, Terao S, Chiba T, Murakami K, Yanaka A, Uehara T, Ishii Y, Soma M, Tajiri H. Adjunct antibiotic combination therapy for steroid-refractory or -dependent ulcerative colitis: an open-label multicentre study. Aliment Pharmacol Ther. 2014 May;39(9):949-56. doi: 10.1111/apt.12688. Epub 2014 Mar 13. PMID 24628398
- [Background] Knoop KA, McDonald KG, Kulkarni DH, Newberry RD. Antibiotics promote inflammation through the translocation of native commensal colonic bacteria. Gut. 2016 Jul;65(7):1100-9. doi: 10.1136/gutjnl-2014-309059. Epub 2015 Jun 4. PMID 26045138